CLINICAL TRIAL: NCT05011253
Title: Electronic Trigger for Microhematuria
Brief Title: Electronic Triggers: Microhematuria Trigger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: QI-MH
Record Dates: First submitted 2021-08-16; First posted 2021-08-18 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Hematuria
MeSH Terms: conditions — Hematuria

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The group which will receive the InBasket message to notify users that a patient has clinically significant microscopic hematuria and makes recommendations for follow-up.
  Interventions: Other: Electronic Trigger Microhematuria Alert
- Control (No Intervention): The group which will not receive the InBasket message to notify users that a patient has clinically significant microscopic hematuria. (Standard practice)

INTERVENTIONS:
Other: Electronic Trigger Microhematuria Alert — To evaluate the effectiveness of an InBasket Results message in prompting providers to place appropriate follow up orders. The message will notify users that a patient has clinically significant microscopic hematuria and is at high risk for underlying malignancy and will include the official recommendations (imaging with a CT urogram, urology evaluation with cystoscopy).
  Arms: Intervention

SUMMARY:
The research team will evaluate the effectiveness of an InBasket Results message that prompts providers to place appropriate follow up orders.

DETAILED DESCRIPTION:
The research team will evaluate the effectiveness of an InBasket Results message that prompts providers to place appropriate follow up orders. The message will notify users that a patient has clinically significant microscopic hematuria and is at high risk for underlying malignancy and will include the official recommendations (imaging with a CT urogram, urology evaluation with cystoscopy).

ELIGIBILITY:
Inclusion Criteria:

* 35 years of age or older
* 3+ RBC on Urinalysis
* Urinalysis sent during an outpatient encounter
* any of the following: 60 years of age or older; RBC > 25; current or prior tobacco use; Gross Hematuria

Exclusion Criteria:

* Under 35 years of age
* Cystoscopy within 1 year prior to Urinalysis
* Nitrite positive AND Leukocyte Esterase positive
* Nitrite positive AND >100 WBC
* Leukocyte Esterase positive AND >100 WBC
* Know GU cancer diagnosis
* Urinalysis ordered by urology provider

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Evaluation rate | 180 days of alert
  Urology evaluation with cystoscopy and appropriate imaging

CONTACTS AND LOCATIONS:
Overall Officials: Saul Blecker, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone, New York, New York, United States